CLINICAL TRIAL: NCT03414281
Title: Transmuscular Quadratus Lumborum Block Versus Thoracic Paravertebral Block for Acute Pain and Quality of Recovery After Laparoscopic Renal Surgery
Brief Title: TMQLB Versus TPVB for Acute Pain and Quality of Recovery After Laparoscopic Renal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: we use this data as a pilot study
Sponsor: Cui Xulei (Other)
Responsible Party: Sponsor-Investigator, Cui Xulei, The attending physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: cuixulei5
Record Dates: First submitted 2018-01-09; First posted 2018-01-29 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Nerve Block, Nephrectomy, Analgesia
Keywords: quadratus lumborum block, thoracic paravertebral block, nephrectomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TMQLB group 1 (Experimental): 0.4ml/kg ropivacaine is injected into the interfascial plane between the psoas major and quadratus lumborum muscle using TMQLB approach.
  Interventions: Procedure: TMQLB group 1
- TMQLB group 2 (Experimental): 0.6ml/kg ropivacaine is injected into the interfascial plane between the psoas major and quadratus lumborum muscle using TMQLB approach.
  Interventions: Procedure: TMQLB group 2
- TPVB group (Active Comparator): 0.4ml/kg ropivacaine is injected into the thoracic paravertebral space (T10) using TPVB approach.
  Interventions: Procedure: TPVB

INTERVENTIONS:
Procedure: TMQLB group 1 — The patient is placed in the lateral position. The curved (C1-5) probe of Philip CX50 Ultrasound Scanner is used for scan and located vertical to the iliac crest at the posterior axillary line to find the Shamrock sign. The 22-G needle is then inserted in plane and directed to the QL muscle. After the proper position of the needle tip between the psoas major muscle and the quadratus lumborum muscle is confirmed, 0. 4 ml/kg 0.5% ropivacaine with 1: 200,000 adrenaline is injected into the interfascial plane.
  Followed by IPCA in the first 48h after surgery: morphine boluses: 1.5-2 mg, lockout time :10 min, 1h limitation: 6-8 mg morphine.
  Arms: TMQLB group 1
Procedure: TMQLB group 2 — The patient is placed in the lateral position. The curved (C1-5) probe of Philip CX50 Ultrasound Scanner is used for scan and located vertical to the iliac crest at the posterior axillary line to find the Shamrock sign. The 22-G needle is then inserted in plane and directed to the QL muscle. After the proper position of the needle tip between the psoas major muscle and the quadratus lumborum muscle is confirmed, 0. 6 ml/kg 0.5% ropivacaine with 1: 200,000 adrenaline is injected into the interfascial plane.
  Followed by IPCA in the first 48h after surgery: morphine boluses: 1.5-2 mg, lockout time :10 min, 1h limitation: 6-8 mg morphine.
  Arms: TMQLB group 2
Procedure: TPVB — The patient is placed in the lateral position, the spinous processes of T10 are identified and marks are made 2cm lateral to the spinous processes. The linear(L12-3) probe of Philips CX50 is placed transversally at the mark to identify the paravertebral space. Then a 22-G needle is inserted in-plane from lateral to medial and advanced until the tip reached the paravertebral space surrounded by the parietal pleura and the superior costotransverse ligament. 0.4 ml/kg 0.5% ropivacaine with 1: 200,000 adrenaline is injected into the paravertebral space of T10.
  Followed by IPCA in the first 48h after surgery: morphine boluses: 1.5-2 mg, lockout time :10 min, 1h limitation: 6-8 mg morphine.
  Arms: TPVB group

SUMMARY:
This trial is a prospective, randomized, single-center, open-label, parallel-arm, blinded-analysis trial, the objective of which is to evaluate the effect of transmuscular quadratus lumborum block (TMQLB) in the pain relief and quality of recovery in laparoscopic renal surgery compared with thoracic paravertebral block (TPVB).

ELIGIBILITY:
Inclusion Criteria:

* 17~80 years of age;
* American Society of Anesthesiologists physical status I-III;
* undergoing laparoscopic nephrectomy.

Exclusion Criteria:

* have a known allergy to the anesthetics being used;
* infection at injection site
* coagulopathy or history of anticoagulants use
* chronic analgesics consumption or history of substance abuse
* inability to properly describe postoperative pain or recovery to investigators (e.g., language barrier, neuropsychiatric disorder).

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
mean VAS of the first postoperative 24 hours | within the first 24 postoperative hours
  VAS is an internationally recognized pain scale with 11 points ranging from 0 to 10 points, with 0 defined as no pain and 10 defined as the worst pain imaginable. The VAS will be registered at 0, 2, 4, 8, 12, 24 hours after the surgery, and the primary outcome will be calculated as the mean VAS scores measured at these time point.

SECONDARY OUTCOMES:
cumulative morphine consumption | at 0, 2,4, 8, 12, 24 ,48, 72hours and 7 day after the surgery
  morphine consumption will be registered at 0, 2, 4, 8, 12, 24, 48, 72 hours and 7 days after the surgery and will be calculated as the sum of the values
long-term pain control | at 48, 72 and 7 days after the surgery
  evaluated by VAS at 48, 72 hours and 7 days after the surgery
dermatomal distribution of sensory loss | 10, 20, 30 and 40 minutes after the intervention
  evaluated at 10, 20, 30 and 40 minutes after the intervention with pinprick test using Von Frey filaments
nausea score | at 0, 2, 4, 8, 12, 24 and 48 hours after the surgery;
pruritus score | at 0, 2, 4, 8, 12, 24 and 48 hours after the surgery;
ambulation time | after the surgery
  time to patient's first walking after the surgery
time of recovery of bowel movement | after the surgery
  defined as the time to first flatus
quality of recovery evaluated by the self-assessment 15-item quality of recovery (QoR) scale | at 3 days and 5 days after the sugery
  QoR is a 15-item questionnaire which will score on a scale of 0-10 pertaining to patient's comfort, support system, pain, well-being, and ability to carry out daily activities, where 0 indicates none of the time and 10 indicates all of the time
postoperative length of hospital stay | after the surgery
  time to patient's discharge
patient satisfaction with anesthesia | at 48 hours after the surgery
  evaluated with the Chinese version of Bauer questionnaire at 48 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Xulei CUI, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan Q, Cui X, Fei Y, Xu Z, Huang Y. Transmuscular quadratus lumborum block versus thoracic paravertebral block for acute pain and quality of recovery after laparoscopic renal surgery: study protocol for a randomized controlled trial. Trials. 2019 May 20;20(1):276. doi: 10.1186/s13063-019-3359-7. PMID 31109368